CLINICAL TRIAL: NCT00718523
Title: A Randomized, Double-blind, Placebo Controlled, Multi-center, Phase II Study of Adding AMG 479, a Fully Human Monoclonal Antibody Against Insulin-like Growth Factor Type 1 Receptor (IGF-1R) to First Line Chemotherapy in Patients With Optimally Debulked ( < 1 cm ) Epithelial Ovarian Cancer
Brief Title: Study of Adding AMG 479 to First Line Chemotherapy in Patients With Optimally Debulked Epithelial Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The steering committee of the TRIO014 study has taken the decision to stop the TRIO014 trial.
Sponsor: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRIO 014
Record Dates: First submitted 2008-07-17; First posted 2008-07-18 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — ganitumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): Placebo plus paclitaxel/carboplatin chemotherapy administered on Day 1 of each 21-day cycle for 6 cycles - then 6 additional cycles of placebo administered on Day 1 of each 21-day cycle.
  Interventions: Drug: AMG 479 Placebo
- B (Experimental): AMG 479 plus paclitaxel/carboplatin chemotherapy administered on Day 1 of each 21-day cycle for 6 cycles - then 6 additional cycles of AMG 479 single agent administered on Day 1 of each 21-day cycle.
  Interventions: Drug: AMG 479

INTERVENTIONS:
Drug: AMG 479 — Solution for infusion - 18 mg/kg on day 1 of each 21-day cycle
  Arms: B
Drug: AMG 479 Placebo — Matching placebo administered Day 1 of each 21 day cycle.
  Arms: A

SUMMARY:
This study will determine the value of adding AMG 479 (fully human monoclonal antibody against IGF-1R) to paclitaxel and carboplatin first line chemotherapy in patients with optimally debulked (<1 cm) FIGO stage III and IV (positive pleural cytology only) ovarian epithelial (including fallopian tube and primary peritoneal) carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed optimally debulked (< 1 cm) FIGO stage III or stage IV (positive pleural cytology only) ovarian epithelial (including fallopian tube and primary peritoneal) carcinoma.
* Patients should have undergone surgical debulking, by a surgeon experienced in the management of ovarian cancer, with the aim of maximal surgical cytoreduction. All patients must be optimally debulked as defined as having no residual tumor of greater than 1 cm in the post surgical setting.
* Patients with stage IV disease will be eligible if a positive pleural cytology is the only extra peritoneal disease.
* Paraffin block (or 10 - 20 unstained slides) and fresh frozen surgical/biopsy specimens of the primary tumor are required at baseline.
* No prior systemic treatment in the primary disease treatment setting.
* Female ≥ 18 years of age or legal age.
* ECOG performance status ≤ 2.
* Adequate organ and bone marrow function
* Non diabetic patients or Type 1 or 2 Diabetic Patients:

  • Diabetes must be controlled with HgbA1c < 8% and fasting blood glucose level <160 mg/dL.
* Patient must be willing and able to comply with scheduled visits, and all study procedures.
* Informed consent obtained.
* Patients should be able to commence systemic therapy within 6 weeks of cytoreductive surgery.
* Life expectancy > 12 weeks.
* Adequate coagulation parameters (within 14 days prior to randomization), International Normalized Ratio (INR) ≤1.5; Activated Prothrombin Time (APTT) ≤ 1.5 x ULN

Exclusion Criteria:

* Non-epithelial ovarian cancer, including malignant mixed Mullerian tumors.
* Borderline tumors (tumors of low malignant potential).
* Planned intraperitoneal cytotoxic chemotherapy.
* Prior systemic anticancer therapy for ovarian cancer.
* Any previous radiotherapy to the abdomen or pelvis.
* Patients with synchronous primary endometrial carcinoma, or a past history of primary endometrial carcinoma, are excluded unless ALL of the following criteria for describing the endometrial carcinoma are met: Stage ≤ Ib, no more than superficial myometrial invasion, no lymphovascular invasion, not poorly differentiated (i.e., not Grade 3 or papillary serous or clear cell).
* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri or curatively treated DCIS/LCIS, or non-melanoma or in situ melanoma skin cancer.
* Prior treatment with a humanized monoclonal antibody anticancer therapeutic.
* Prior treatment with investigational treatment targeted to IGF axis including, but not limited to, CP 751,871, IM-A12, RO4858696.
* Previous exposure to AMG 479.
* Anticipation of a need for a major surgical procedure or radiation therapy during the study.
* History of hypersensitivity to recombinant proteins.
* Treatment with radiotherapy, surgery, or an investigational agent within 4 weeks of randomization.
* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, cerebrovascular accident or transient ischemic attack, grade > 2 peripheral neuropathy, pulmonary embolism, deep vein thrombosis, or other thromboembolic event.
* History of brain metastases, spinal cord compression, or carcinomatous meningitis.
* Patient of child-bearing potential is pregnant (eg, positive human chorionic gonadotropin test) or is breast feeding.
* Patient of child-bearing potential is not willing to use adequate contraceptive precautions.
* Known active infection, or on antiretroviral therapy for HIV disease.
* Known positive test for chronic hepatitis B or C infection.
* Any other underlying physical or mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
* Refusal or inability to give informed consent to participate in the study.
* Other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the patient's safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried E Konecny, MD, Study Chair — University of California, Los Angeles
Locations (55):
- United States (23):
  - Central Hematology Oncology Medical Group Inc., Alhambra, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - St Jude Heritage Healthcare, Fullerton, California
  - Wilshire Oncology Medical Group Inc, La Verne, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - University of California San Francisco, San Francisco, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Memorial Cancer Institute, Hollywood, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute Emory University School of Medicine, Atlanta, Georgia
  - Hematology and Oncology Specialists, LLC, Metairie, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Toledo Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - London Health Science Center, London, Ontario
  - CHUM Hopital Notre Dame, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- France (4):
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Centre Léon Bérard, Lyon
  - Clinique Hartmann, Neuilly-sur-Seine
  - Institut Curie, Paris
- Germany (9):
  - Charite Campus Benjamin Franklin, Berlin
  - University Hospital Charite, Berlin
  - Universitat Bonn, Bonn
  - Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Universitatsklinikum des Saarlandes, Homburg
  - Klinikum Kassel, Kassel
  - Rotkreuzkrankenhaus Munchen, Munich
  - Universitats Frauenklinik Tubingen, Tübingen
- Ireland (2):
  - St Jame's Hospital, Dublin
  - Waterford Regional Hospital, Waterford
- Israel (5):
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - Asaf Harofe MC, Zrifin
- Spain (5):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital U 12 de Octubre, Madrid
  - Hospital Universitario de Tenerife, San Cristóbal de La Laguna
  - Hospital Universitario Virgen Macarena de Sevilla, Seville
- United Kingdom (3):
  - Saint James's University Hospital, Leeds
  - University College London, London
  - Mount Vernon cancer centre, Northwood

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted over a total of 55 sites in 8 countries.
Groups:
- A Control: Placebo plus paclitaxel/carboplatin chemotherapy administered on Day 1 of each 21-day cycle for 6 cycles - then 6 additional cycles of placebo administered on Day 1 of each 21-day cycle.
  AMG 479 Placebo: Matching placebo administered Day 1 of each 21 day cycle.
- B Experimental: AMG 479 plus paclitaxel/carboplatin chemotherapy administered on Day 1 of each 21-day cycle for 6 cycles - then 6 additional cycles of AMG 479 single agent administered on Day 1 of each 21-day cycle.
  AMG 479: Solution for infusion - 18 mg/kg on day 1 of each 21-day cycle
Period: Overall Study
Arm/Group | A Control | B Experimental
Started | 84 | 86
Completed | 66 | 62
Not Completed | 18 | 24
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Death | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Control | B Experimental | Total
Number analyzed (Participants) | 84 | 86 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 61 | 120
  >=65 years | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.0) | 57.2 (12.3) | 57.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 86 | 170
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 34 | 59
  United Kingdom | 1 | 2 | 3
  Canada | 4 | 6 | 10
  France | 7 | 3 | 10
  Israel | 2 | 2 | 4
  Spain | 1 | 1 | 2
  Germany | 44 | 38 | 82
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Number; unit: participants] — 6-point (0 to 5) ordinal scale to assess how the disease affects the daily living abilities of the patients and determine appropriate treatment and prognosis
  participants
    PS 0 (fully active) | 36 | 32 | 68
    PS 1 (restricted in physically strenuous activity) | 43 | 46 | 89
    PS2(ambulatory and capable of all selfcare) | 5 | 6 | 11
    Missing | 0 | 2 | 2
Time from Surgery to first treatment dose [Mean (Standard Deviation); unit: weeks] | 5.1 (1.2) | 5.1 (1.4) | 5.1 (1.3)
Time from diagnosis to randomization [Mean (Standard Deviation); unit: weeks] | 5.2 (2.3) | 5.4 (3.4) | 5.3 (2.9)
Origin of tumor [Number; unit: participants]
  Primary peritoneal | 8 | 4 | 12
  Fallopian tube | 4 | 4 | 8
  Ovarian | 69 | 77 | 146
  Ovarian + Primary peritoneal | 0 | 1 | 1
  Ovarian + Fallopian tube | 2 | 0 | 2
  Missing | 1 | 0 | 1
Stage at first diagnosis (International Federation of Gynecology and Obstetrics (FIGO)) [Number; unit: participants] — 5-point ordinal scale to assess the extent of the disease (0->IV). Roman numeral staging from the less to the most advanced cancer. Individual stage (I to III) is broken down in substage: IA, IB, IC,...
  participants
    IIIA | 3 | 2 | 5
    IIIB | 10 | 6 | 16
    IIIC | 65 | 72 | 137
    IV | 6 | 6 | 12
Histopathologic type [Number; unit: participants]
  papillary serous | 69 | 72 | 141
  mucinous | 0 | 1 | 1
  endometroid | 4 | 5 | 9
  clear cell | 2 | 2 | 4
  mixed | 5 | 3 | 8
  other | 4 | 3 | 7
Histologic Grade [Number; unit: participants] — Cancer cells compared with normal cells
  participants
    G1 (well differentiated) | 1 | 5 | 6
    G2 (moderately differentiated) | 15 | 18 | 33
    G3 (poorly differentiated) | 65 | 57 | 122
    Not done | 3 | 6 | 9
Number of prior therapies [Number; unit: participants] — Prior anti-tumor treatment characteristics
  participants
    1 therapy | 80 | 78 | 158
    2 therapies | 4 | 8 | 12
CA 125 status [Number; unit: participants]
  with elevated CA 125 | 67 | 70 | 137
  with CA 125 in the normal range | 17 | 15 | 32
  missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS): Time From Randomization Until Date of Progression or Death.
Description: A patient may have been declared to have progressive disease on the basis of radiological measuremt of tumor lesions assessmt or CA125 evaluation (tumor measuremts taking precedence).Radiological progression was defined as per the RECIST guidelines (Therasse et al, JNCI2000) as at least 20% increase in the sum of the longest diameters of target lesions(ref the smallest sum of the longest diam recorded since the treatmt started or since the appearance of at least 1 new lesion).Serum CA125 progression was defined, according to the 2005 GCIG def: pts with:
  * Elevated CA125 pretreatmt and normalization of CA125 has to show evidence of CA125≥ 2 times the upper normal limit on 2 occasions at least 1 wk apart OR
  * Elevated CA125 pretreatmt which never normalized must show evidence of CA125≥ 2 times the nadir value on 2 occasions at least 1 wk apart OR
  * CA125 in the normal range pretreatmt had to show evidence of CA125 ≥ 2 times the upper normal limit on 2 occasions at least 1 wk apart
Time Frame: Radiological tumor assessment: every 12(+/- 1) weeks for 3 years after randomization + CA 125: day 1 of each cycle
Population: Unstratified Intent To Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A Control | B Experimental
Number analyzed (Participants) | 84 | 86
months | 16.690 [14.686 to 28.123] | 15.737 [12.090 to 21.388]

2. Secondary Outcome: Time To Progression (TTP): Interval From the Date of Randomization to the Date of Disease Progression
Description: as for outcome 1
Time Frame: Radiological tumor assessment: every 12 (+/- 1) weeks for 3 years after randomization + CA125: day 1 of each cycle
Population: Unstratified Intent To Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A Control | B Experimental
Number analyzed (Participants) | 84 | 86
months | 17.840 [14.784 to 34.037] | 16.066 [12.090 to 22.341]

3. Secondary Outcome: Overall Survival (OS)
Description: Interval between the date from randomization to death from any cause whichever came first.
Time Frame: Day 1 of each cycle up to 4 years after randomization
Population: Unstratified Intent To Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A Control | B Experimental
Number analyzed (Participants) | 84 | 86
months | NA [NA to NA] — The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time. | 45.207 [45.207 to NA] — The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.

ADVERSE EVENTS:
Time Frame: The monitoring period for AEs started from signature of the ICF and continued up to 30 days after last dose.
Description: For participant flow module it is based on Intent To Treat so the patients are counted according to their "randomization group".For "participants at risk" the patients are grouped by the "actual treatment" 4 patients were allocated with incorrect treatment and received AMG479 instead of Placebo.The total number of patients treated remains the same.
Arm/Group | A Control | B Experimental
Serious Adverse Events (participants affected / at risk) | 31/77 | 30/88
Other Adverse Events (participants affected / at risk) | 77/77 | 86/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Control (N=77) | B Experimental (N=88)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 5 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
General Physical health deterioration (General disorders) | 1 (1) | 5 (5)
non cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 3 (3)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 2 (4) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes melitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Control (N=77) | B Experimental (N=88)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 8 (8)
Vision blurred (Eye disorders) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 28 (33) | 28 (32)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 11 (13)
Stomatitis (Gastrointestinal disorders) | 17 (19) | 24 (25)
Chills (General disorders) | 4 (4) | 10 (12)
Fatigue (General disorders) | 46 (55) | 49 (55)
Oedema peripheral (General disorders) | 8 (8) | 5 (5)
Pain (General disorders) | 9 (10) | 11 (11)
Pyrexia (General disorders) | 13 (15) | 9 (12)
Hypersensitivity (Immune system disorders) | 10 (14) | 8 (10)
Bronchitis (Infections and infestations) | 5 (5) | 2 (2)
Cystitis (Infections and infestations) | 5 (9) | 2 (2)
Nasopharyngitis (Infections and infestations) | 12 (13) | 7 (10)
Weight increased (Investigations) | 2 (2) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 16 (17) | 12 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 8 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (26) | 27 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (17) | 11 (13)
Dysgueusia (Nervous system disorders) | 15 (17) | 15 (16)
Headache (Nervous system disorders) | 17 (20) | 23 (30)
Neuropathy peripheral (Nervous system disorders) | 15 (17) | 24 (25)
Paraesthesia (Nervous system disorders) | 7 (9) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 32 (35) | 27 (31)
Polyneuropathy (Nervous system disorders) | 11 (11) | 8 (8)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 6 (6) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 68 (68) | 66 (66)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (15) | 11 (12)
Hot flush (Vascular disorders) | 13 (13) | 7 (8)
Hypertension (Vascular disorders) | 3 (3) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 16 (16) | 18 (22)
Abdominal Pain Upper (Gastrointestinal disorders) | 14 (16) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 24 (32) | 37 (45)
Nausea (Gastrointestinal disorders) | 51 (67) | 46 (53)
Vomiting (Gastrointestinal disorders) | 31 (38) | 29 (32)
Asthenia (General disorders) | 9 (17) | 5 (6)
Urinary Tract Infection (Infections and infestations) | 11 (15) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (39) | 30 (34)
Bone Pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 18 (21)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 15 (16) | 9 (9)
Syncope (Nervous system disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 12 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 12 (13)
Rash (Skin and subcutaneous tissue disorders) | 17 (22) | 24 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No